CLINICAL TRIAL: NCT01618513
Title: Treatment of Acromegaly With Somatostatin Analogs: GH vs. IGF-I as Primary Biochemical Target
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other); Herlev Hospital (Other); Copenhagen University Hospital, Denmark (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOM-2012-01
Record Dates: First submitted 2012-06-04; First posted 2012-06-13 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2014-12

CONDITIONS: Acromegaly
Keywords: Acromegaly; Somatostatin analogs; Treatment
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SA monitored by GH (Experimental)
  Interventions: Drug: Sandostatin® LAR
- SA monitored by IGF-I (Experimental)
  Interventions: Drug: Sandostatin® LAR
- Control (No Intervention): Control, patients who have achieved sufficient disease control by surgery alone.

INTERVENTIONS:
Drug: Sandostatin® LAR — Intramuscular injections, dosage based on either GH or IGF-I levels.
  Arms: SA monitored by GH; SA monitored by IGF-I

SUMMARY:
Treatment of acromegaly with somatostatin analogs (SA) is well-established and are primarily used after insufficient surgical intervention, but also as primary medical treatment in selected patients. Evaluation of treatment control is based on monitoring blood levels of growth hormone (GH) and insulin-like growth factor-I (IGF-I). However, evaluation of disease control during SA treatment is not always straightforward. It is usually based on normalization of IGF-I and achievement of a certain GH level. In approximately 40% of patients discordant values of GH and IGF-I levels are seen after treatment with SA, with normalized IGF-I levels, despite elevated GH levels. The mechanism behind this observation is unknown, but it indicates that SA may affect this difference.

The primary objective of this study is to investigate if disease control during SA treatment is best achieved by monitoring either GH or IGF-I.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 18 years
* Capable and of age
* Diagnosed with acromegaly
* Sufficient treated for at least 6 months prior to enrollment

Exclusion Criteria:

* Pregnancy or nursing
* Any disease that may compromise the ability to comply with the protocol, as assessed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life | Baseline and after 12 months
  AcroQol (Acromegaly Quality of Life Questionnaire) and PASQ (Patient-Assessed Acromegaly Symptom Questionnaire)

SECONDARY OUTCOMES:
SA dosage | After 12 months of treatment
  SA dosage at last follow-up
Change in glucose, FFA and insulin | Baseline and after 12 months
  Glucose tolerance during an oral glucose load of 75 gram of glucose
Change in discordant GH/IGF-I levels | Baseline and after 12 months
  Discordant GH/IGF-I levels are recorded.
New biomarkers of treatment evaluation | Baseline and after 12 months
  New biomarkers of GH/IGF-I status (bioactive IGF-I)
New biomarkers of treatment evaluation2 | Baseline and after 12 months
  New biomarkers of GH/IGF-I status (free GH)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L. Jørgensen, Professor, Study Chair — Aarhus University Hospital
Locations (1):
- Department of Endocrinology, Aarhus University Hospital, Aarhus C, Denmark